# **Title:**

Effect of Pomegranate Seed Powder on

markers of Metabolic Syndrome

# NCT:

Not Assigned yet

# **Submission Date:**

Uploaded here on 21st June, 2023

## **STATEMENT OF PROBLEM**

A number of chronic disorders can lead to metabolic syndrome, which has been identified as one of the key risk factors for the epidemic of type 2 diabetes and cardiovascular diseases in the twenty-first century. Thus, it's a high time to mitigate the prevalence of these risk factors to overcome metabolic syndrome.

## **Objective:**

To evaluate the effectiveness of pomegranate seed powder supplementation in preventing metabolic dysfunction and its main risk factors, such as hypertension and cardiovascular illnesses.

### **Study Protocol**

## **Type of Study**

This trail is prospective clinical type.

#### **Supplement preparation**

Pomegranate seeds and arils will be separated, and then the seeds will be dried for 15 days in a lab environment. Later, a mechanical grinder will be used to powder the dried seeds. PS powder (PSP) will be packed in a capsule form, 5 g in each.

## **Participants**

The population under study will be consisted of people suffering with any of the three metabolic impairments; Insulin resistance, obesity, disturbed glucose level, hyper-cholesterol, hypertension and higher blood pressure. Exclusion criteria will be critically ill or hospitalized patients and individuals with digestion and absorption issues.

#### Span of study

The clinical trial on the 50 patients of metabolic syndrome will be conducted for the duration of 8 weeks with the supplementation of PSP capsule, twice a day.

#### **Outcome Evaluation**

Blood pressure, total cholesterol, and triglycerides (TG) will be measured at the enrollment point (i.e., baseline) and at the end of the 8-week intervention period. Fasting blood glucose (FBG), glycated haemoglobin (HbA1c), and triglycerides (TG) will be measured at the enrollment point (i.e., baseline). A fresh blood sample from a vein will then be taken and examined. A calibrated digital weight scale will also be used to check the patient's weight. Detail of all data collected is as follows:

### **Anthropometric Measurements:**

- Weight
- Height
- Skin fold Thickness

#### **Biochemical Evaluation:**

- Blood Pressure
- Fasting Blood Glucose
- Total Cholesterol
- Triglycerides

#### **Clinical Evaluation:**

Obesity

### **Statistical Analysis Plan**

Using one-way ANOVA, the statistical significance of the host parameter data will be determined (SPSS Inc., Chicago, IL, USA). When the p-values are less than 0.05, differences are considered significant. Statistical analyses will be carried out in the R programming environment for data sequencing. For both quantitative and qualitative variables, data will be displayed as  $\pm$  SD or frequency (percent), respectively.